CLINICAL TRIAL: NCT06142409
Title: The Effect of Non-biocidal Adjuncts on the Formation, Composition, Functionality, and Microscale Architecture of Dental Biofilms: a Randomized Controlled Trial
Brief Title: Effect of Enzyme-containing Lozenge on Dental Biofilm Formation, Composition and Functionality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novozymes A/S (Industry)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NZ-2022-05
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Dental Biofilm Accumulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Active Comparator): Enzyme-containing lozenge
  Interventions: Dietary Supplement: Enzyme containing lozenge
- Placebo arm (Placebo Comparator): Placebo lozenge
  Interventions: Dietary Supplement: Enzyme containing lozenge

INTERVENTIONS:
Dietary Supplement: Enzyme containing lozenge — Lozenge containing multiple enzyme combination

SUMMARY:
A double-blind, placebo-controlled randomized cross-over trial evaluating the effect of enzyme-containing lozenge on in vivo and in situ grown dental biofilm accumulation. The study includes two phases, one each for the investigation of in-vivo and in-situ grown dental biofilm

DETAILED DESCRIPTION:
Up to 50 subjects (aged ≥ 18 years old) with 3 or more active caries lesion, will be randomized to receive:

Phase 1: The effect of multiple-enzyme treatment on plaque accumulation in vivo

Phase 1 includes two experimental periods lasting for one day each, with a washout period of two weeks in between. Each experimental period will include two visits, at day 0 and day 1.

At day 0, the participants will receive a professional tooth cleaning and be randomized to receive Sequence 1 or Sequence 2 in a double-blind randomized cross-over design:

Sequence 1: 3 active enzyme-containing lozenges per day for one day (app. 24h) followed by a washout period of two weeks, followed by 3 identical placebo lozenges per day for one day (app. 24h).

Sequence 2: 3 placebo lozenges per day for one day (app. 24h) followed by a washout period of two weeks, followed by 3 identical active enzyme lozenges per day for one day (app. 24h).

The participants will be instructed to take one lozenge three times (morning, noon, evening) for one day. No normal oral hygiene procedures will be allowed during the intervention periods of one day. At the end of both experimental phases, plaque is assessed using planimetric recordings obtained with an intraoral camera and TM-QHPI to provide information on the individual level of plaque formation.

Phase 2: The effect of multiple-enzyme treatment on in situ-grown biofilms

The phase is designed in a double-blind randomized cross-over design, including two experimental periods lasting for 2 days, with a washout period of 5 days in between. Each experimental period will include two visits, on day 0 and day 2. Oral biofilms will be grown in situ on prefabricated non-fluorescent glass slabs for 48 hours. The glass slabs will be mounted on the individual lower-jaw splints.

At day 0, the participants will be randomized to receive Sequence 1 or Sequence 2:

Sequence 1: 3 active enzyme-containing lozenges per day for 2 days followed by a washout period of 5 days, followed by 3 identical placebo lozenges per day for 2 days.

Sequence 2: 3 placebo lozenges per day for 2 days followed by a washout period of 5 days, followed by 3 identical active enzyme lozenges per day for 2 days.

Oral biofilms will be grown in situ on prefabricated non-fluorescent glass slabs for 2-4 experimental periods of 48 hours. After each experimental period, the in situ-grown biofilms will be collected and stored in a research biobank.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years old.
* Have three or more active carious lesions.
* Anatomically possible to manufacture an intraoral lower-jaw splint.
* Able to understand and follow instructions, as well as to read and sign the informed consent form.
* A plaque index score ≥ 2 according to the Turesky Modification of the Quigley-Hein Plaque Index (TM-QHPI), following 8 to 12 hours plaque accumulation period.

Exclusion Criteria:

* History of allergies towards any of the ingredients in the test products
* Self-reported pregnant or nursing
* Antibiotic or anti-inflammatory medication within 90 days of the screening visit.
* Orthodontic appliances, including retainers, or removable partial dentures.
* Self-reported serious medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Change in in-vivo dental biofilm accumulation | 1 day
  To investigate the effect of an enzyme-containing lozenge on dental biofilm accumulation in caries-active subjects in vivo assessed by the planimetric plaque index (PPI)

SECONDARY OUTCOMES:
Change in in-vivo dental biofilm accumulation | 1 days
  To investigate the effect of an enzyme-containing lozenge on dental biofilm accumulation in caries-active subjects in vivo assessed by the Turesky-modified Quigley Hein Plaque Index (TM-QHPI)
Change in in-situ grown dental biofilm accumulation | 2 days
  The effect of enzyme-containing lozenge on changes in the microarchitecture of in situ-grown biofilms from caries-active subjects analyzed by optical coherence tomography.
Change in oral microbial community composition of in-situ grown dental biofilm | 2 days
  Shift in oral microbial community composition of in situ-grown biofilms from caries-active subjects assessed by next-generation sequencing of 16S rRNA genes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dentistry and Oral Health, Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No